CLINICAL TRIAL: NCT03457519
Title: Children's Automated Respiration Monitor (ChARM) for Child Pneumonia Diagnosis by Community Health Workers in Mali: Innovating ChARM's Role in Supervision, Training and Diagnosis, a Cluster Randomized Control Trial
Brief Title: Children's Automated Respiration Monitor (ChARM) for Child Pneumonia Diagnosis by Community Health Workers in Mali
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diego Bassani (Other)
Collaborators: Canadian Red Cross (Other)
Responsible Party: Sponsor-Investigator, Diego Bassani, Director, International Program Evaluation Unit (IPE), Center for Global Child Health, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R-ST-POC-1707-07682
Record Dates: First submitted 2017-12-14; First posted 2018-03-07 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Acute Respiratory Infection
Keywords: ChARM; community health worker

STUDY DESIGN:
Intervention Model Description: Intervention Group A - Community Health Workers (CHWs) (Basic training in CHW curriculum, ChARM training and 8-month application of the ChARM device, self-monitoring, direct observation and review of CHW routine monthly reports and drug supply sheets): 8 months, March- November 2018.
  Intervention Group B - Community Health Workers (Basic training in CHW curriculum, ChARM training and 4-month application of the ChARM device, self-monitoring, direct observation and review of CHW routine monthly reports and drug supply sheets): March- November 2018.
  Control Group C - Community Health Workers (Basic training in CHW curriculum, direct observation and CHW routine monthly reports and drug supply sheets): 8 months, March- November 2018.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group A (Active Comparator): CHWs trained in ChARM and using ChARM as a self-monitoring tool for 8 months while counting respiratory rate of children under 5 visually using a timer.
  Intervention: The Children's Respiration Monitor (also known as ChARM) device is routinely used to diagnose Pneumonia cases but in this study it will be used as a self-monitoring and teaching aide for strengthening CHWs skills.
  Interventions: Device: Children's Automated Respiration Monitor (ChARM)
- Intervention Group B (Active Comparator): CHWs trained in ChARM and using ChARM as a self-monitoring tool for 4 months while counting respiratory rate of children under 5 visually using a time; then discontinue using ChARM and continue to monitor the respiratory rate visually using a timer only for the remaining 4 months.
  Intervention: The Children's Respiration Monitor (also known as ChARM) device is routinely used to diagnose Pneumonia cases but in this study it will be used as a self-monitoring and teaching aide for strengthening CHWs skills.
  Interventions: Device: Children's Automated Respiration Monitor (ChARM)
- Control Group C (No Intervention): CHWs who did not receive the ChARM training and will be monitoring the respiratory rate of children under 5 visually using a timer only, as per the MoH traditional training.

INTERVENTIONS:
Device: Children's Automated Respiration Monitor (ChARM) — The Philips CHARM (children's automatic respiratory monitor) is specifically designed to detect pneumonia in low resource areas. The lightweight measuring device sits on a child's or infant's chest, secured by a strap and measures respiration rate (fast breathing) through an ingenious algorithm. In this study ChARM will be used as a self monitoring and teaching aide by the CHWS.
  Arms: Intervention Group A; Intervention Group B

SUMMARY:
The primary objective of this study is to estimate the impact of a self-monitoring tool (ChARM), used as a teaching/monitoring device, on the CHWs respiratory rate counting accuracy when assessing children under the age of 5 years with suspected pneumonia symptoms.

DETAILED DESCRIPTION:
Methodology:

The study is designed as a community based, cluster randomized, pragmatic, intervention trial. It will be conducted within the existing 2016-2020 project structure. Specifically, the intervention will evaluate the potential of the ChARM device to improve CHWs competency in counting respiratory rate and diagnose pneumonia more accurately in children under 5 years presenting with symptoms in remote areas.

Intervention Group A - Community Health Workers (CHWs) (Basic training in CHW curriculum, ChARM training and 8-month application of the ChARM device, self-monitoring, direct observation and review of CHW routine monthly reports and drug supply sheets): 8 months, March- November 2018.

Intervention Group B - Community Health Workers (Basic training in CHW curriculum, ChARM training and 4-month application of the ChARM device, self-monitoring, direct observation and review of CHW routine monthly reports and drug supply sheets): 8 months,March- November 2018.

Control Group C - Community Health Workers (Basic training in CHW curriculum, direct observation and CHW routine monthly reports and drug supply sheets): 8 months, March- November 2018.

CHW and Field Monitor In-depth interviews - November 2018

Data analysis and report writing - December 2018-January 2019

ELIGIBILITY:
Inclusion Criteria:

* • Be currently providing iCCM services on a full-time basis to the populations they are serving.

  * Have completed the Malian Ministry of Health basic community health care worker training provided as part of the 2016-2020 Strengthening Maternal, Newborn and Child Health project.
  * Are using a device (a respiratory timer) as part of their basic MoH training package, or have a cell phone to use to count the respiratory rates of children under five with suspected symptoms of pneumonia.
  * Be willing to participate in a trial to study the impact of using ChARM as a self-monitoring tool to improve the capacity to detect pneumonia.

Exclusion Criteria:

* • CHWs in conflict ridden geographical areas within the district or not, providing consistent services on a full-time basis to the populations they are serving.

  * CHWs not willing to participate in the trial.
  * CHWs who do not have a device (watch, respiratory timer or cell phone) to support measurement of respiratory rates and who are not routinely counting respiratory rate to diagnose suspected pneumonia.
  * CHWs who did not complete the MoH basic training for CHWs provided through the 2016-2020 Strengthening Maternal, Newborn and Child Health program

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Acute Respiratory Illness (ARI) Case fatality rate | 8 months
  Acute Respiratory Illness (ARI) Case fatality rate defined as number of deaths from respiratory infections among children diagnosed with respiratory infections

SECONDARY OUTCOMES:
Respiratory rate counting accuracy | 8 months
  Respiratory rate is defined as the number of breaths taken per minute
Proportion of pneumonia cases detected and treated by CHWs | 8 months
  Proportion of pneumonia cases detected by the CHWs that are treated by CHWs
Proportion of suspected severe pneumonia cases referred by CHWs to the CSCom | 8 months
  Proportion of all suspected severe pneumonia cases identified by the CHWs (based on presence of fever and increased respiratory rates for age) referred by CHWs to the CSCom
Proportion of suspected pneumonia cases in the community who sought care from a CHW | 8 months
  Proportion of self-referenced pneumonia cases in the community (via household survey) who report seeking care from a CHW
Accuracy in drug management and procurement requests | 8 months
  Percent of CHW with no stock-outs in the last 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Diego G Bassani, PhD, Principal Investigator — University of Toronto
Locations (2):
- Mali (2):
  - iCCM sites, Banamba, Koulikoro
  - iCCM Sites, Koulikoro

IPD SHARING:
Plan to Share IPD: Yes
Plan to share Study Protocol and Clinical Study Reports with local study partners with the purposes of future decisions on future CHW training
Supporting Information: Study Protocol, CSR
Time Frame: March 2018 - March 2019
Access Criteria: Study Protocol and Clinical Study Reports will be shared with local partners - Mali Red Cross, Canadian Red Cross and Mali Ministry of Health

DOCUMENTS (1):
  • Study Protocol (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03457519/Prot_001.pdf